CLINICAL TRIAL: NCT05791890
Title: Observational Study on the Incidence of Infections in Patients With Relapsed/Refractory FMS-like Tyrosine Kinase 3 Acute Myeloid Leukemia Treated With Gilteritinib
Brief Title: GilteRInf 2022 Study (Gilteritinib Related Infections)
Acronym: GilteRInf
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Maria Ilaria Del Principe, Associate Professor, University of Rome Tor Vergata
Other Study IDs: GilteRInf 2022
Record Dates: First submitted 2023-03-05; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: relapsed/refractory acute myeloid leukemia; FLT3+; FLT3 inhibitors; Gilteritinib; infections
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Infections | interventions — gilteritinib

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who receive or have received Gilteritinib: the retrospective part, clinical data will be collected on all patients with LMA FLT3+ (ITD or TKD mutation) treated with Gilteritinib from when the drug was approved and marketed in Italy (April 2, 2020) until April 30, 2022. Enrollment in the prospective cohort will have an estimated duration of 24 months from the time of study approval.
  Interventions: Drug: Gilteritinib
- Case control: for each case of a patient receiving salvage monotherapy with Gilteritinib, a control patient with R/R AML FLT3+ on salvage chemotherapy should also be included.
  Interventions: Drug: Gilteritinib

INTERVENTIONS:
Drug: Gilteritinib — observational study to evaluate the incidence of infections during therapy with Gilteritinb

SUMMARY:
The study is observational, retrospective-prospective, multicenter "real-life" study involving 26 centers belonging to the SEIFEM group. The goal of this study is to obtain a real-life experience in the management and outcome of infectious issues of patients with relapsed/resistant acute myeloid leukemia who receive Gilteritinib therapy, given that recent approval of this drug.

DETAILED DESCRIPTION:
The study is observational, retrospective-prospective, multicenter "real-life" study. Regarding the retrospective part, clinical data will be collected on all patients with acute myeloid leukemia FLT3+ treated with Gilteritinib from when the drug was approved and marketed in Italy (April 2, 2020) until April 30, 2022. Enrollment in the prospective cohort will have an estimated duration of 24 months from the time of study approval. Patients enrolled in the last month will be followed for six months from the date of enrollment to check for the occurrence of any infections. For each case of a patient receiving salvage monotherapy with Gilteritinib, a control patient with relapsed/refractory FLT3+ acute myeloid leukemia on salvage chemotherapy should also be included.

ELIGIBILITY:
Inclusion Criteria:

Population

* All patients with FLT3+ relapsed/refractory AML to any line of therapy treated with Gilteritinib
* Patients ≥18 years of age
* Signature of appropriate informed consent

Exclusion criteria:

- Patients < 18 years old

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Relapsed/refractory AML patients
Sampling Method: Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
absolute infectious risk in patients treated with Gilteritinib, Infection events of grade 3 or more ( CTCAE v.5.0 ) | 24 months
  To assess "real-life" in patients with relapsed/refractory FLT3+ LMA treated with Gilteritinib the absolute infectious risk and compare it with relapsed/refractory patients receiving chemotherapy. The

CONTACTS AND LOCATIONS:
Overall Officials: Maria Ilaria Del Principe, Prof, Principal Investigator — University of Rome Tor Vergata
Locations (1):
- Maria Ilaria Del Principe, Roma, RM, Italy

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/90/NCT05791890/Prot_SAP_000.pdf